CLINICAL TRIAL: NCT06467240
Title: Evaluation of the Hybrid Rapid Maxillary Expander Assisted With Micro-osteo Perforation (MOPs) in Adults: A Prospective Clinical Study
Brief Title: Evaluation of the Hybrid Rapid Maxillary Expander Assisted With Micro-osteo Perforation (MOPs) in Adult.
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ellamey, Principal Investigator, Al-Azhar University
Other Study IDs: 984/3700
Record Dates: First submitted 2024-05-19; First posted 2024-06-20 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Maxillary Anomaly
Keywords: maxillary expansion; Micro-osteo perforation; Cross Bite
MeSH Terms: conditions — Malocclusion | interventions — morpholinopropane sulfonic acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- intervention group: will receive a hybrid rapid maxillary expander assisted by Micro-osteo perforation (MOPs) in mid palatine suture
  Interventions: Procedure: hybrid rapid maxillary expander assisted with Micro-osteo perforation (MOPs)
- control group: will receive a hybrid rapid maxillary expander without any thing
  Interventions: Procedure: hybrid rapid maxillary expander assisted with Micro-osteo perforation (MOPs)

INTERVENTIONS:
Procedure: hybrid rapid maxillary expander assisted with Micro-osteo perforation (MOPs) — patients with constricted maxillary will applied for hybrid expansion and group of them will assisted by Micro-osteo perforation (MOPs)

SUMMARY:
This study will be directed for Evaluation of the hybrid rapid maxillary expander assisted with Micro-osteo perforation (MOPs) in adults

DETAILED DESCRIPTION:
Transverse maxillary deficiencies are common orthodontic issues observed by professionals. It is estimated that 9.4% of adult orthodontic patients have a transverse maxillary deficiency in combination with a posterior cross bite. A normal transverse skeletal relationship between basal bones is fundamental to achieving a satisfactory and stable occlusion.

Therefore, to correct a maxillary transverse deficiency, palatal expanders are needed. Since Haas popularized this technique in the early 1960s, rapid palatal expanders are the most popular devices of choice, characterized by safety, predictability and efficiency.

The rapid process of activation reduces dental movements (side effects) thus enabling skeletal expansion. Surprisingly, only 30% of the expander opening seems to result in suture opening, whereas one-third reflects alveolar bending and another 30% dental movement.

During activations of traditional tooth-borne rapid palatal expansion devices, heavy transverse forces are generated in a short period of time, causing disruption of the inter sutural tissue thus producing midpalatal suture opening.

On many occasions, these expansion forces in-vivo are in the range of 75-120 N, measured at the level of the hyrax screw of the connecting stainless-steel wire arms at the buccal crowns. In vitro skeletal hybrid expanders, before plastic deformation, demonstrated expansion force values from 67 ± 13 N to 183 ± 48 N when tested on the mini-implant's reinforced bone-anchored wire arms .With these forces, the opening of the palatal suture in adolescents or young adults can be frequently unsuccessful.

Therefore, conventional expanders, under high loads, deform prematurely or create excessive molar tipping or mucosa soreness before

reaching midpalatal suture opening. If these expansion forces are not able to open the suture, surgically assisted rapid palatal expansion (SARPE) is suggested.

In addition, scientific papers do not provide information of the amount of force at the level of the midpalatal suture and the limit of plastic deformation. Solely anchored on orthodontic mini-implants (OMIs) and placed in the anterior-middle palate. These bone anchored expanders seem to improve the aforementioned drawbacks and provide greater expansion forces to facilitate midpalatal suture opening even in adult patients so as to avoid SARPE.

Major areas of resistance to hybrid rapid maxillary expansion are mid palatine suture and the pterygomaxillary articulation. With increasing the age, the interdigitation at sutures increases making the site more rigid. The concept of regional acceleratory phenomenon (RAP) can be used for such clinical challenges by using mild surgical trauma induced by Micro-osteo perforation (MOPs) to produce localized inflammation with the mid palatine suture being the only sight easily accessible for intervention, minimally invasive procedures like Micro-osteo perforation (MOPs) can be used to disrupt the mid palatine suture to make it more pliable to expansion forces.

Micro-osteo perforation (MOPs) along the mid palatal suture which will induce rapid acceleratory phenomenon which would accelerate the bone turnover and reduce the regional bone density leading to transient osteopenia and thus bringing out changes in the transverse dimension.

Cone beam computed tomography (CBCT) allows better imaging at low radiation dosages and presents a clear view of bony structures, tooth position, and type of palatal suture fusion with minimal image distortion. Although hybrid rapid maxillary expansion and minimally

invasive surgical techniques are often used in orthodontic clinical practice, only a few studies have been published in the literature on large groups of patients that present possible complications that may occur after practicing this method of orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* An age range from 17-23 years.
* Transverse maxillary deficiency.
* Maxillary lingual Cross bite (unilateral or bilateral)
* No history of previous orthodontic treatment.
* Good oral and general health.
* No systemic condition that could interfere with orthodontic treatment.

Exclusion Criteria:

* Patient with craniofacial anomalies .
* History of extraction of permanent teeth.
* Previous orthodontic treatment.
* Poor oral hygiene or periodontally compromised patient.
* Previous history of bruxism, trauma or par functions.

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: randamly selected
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
CBCT measurment | 3 weeks
  amount of skeletal and dental expansion
suture opening | 3 weeks
  amount of skeletal and dental expansion

CONTACTS AND LOCATIONS:
Overall Officials: Raafat El ghetany Mohamed, professor, Study Director — Al-Azhar University; Ahmed Akram El-Awady, Lecturer, Study Director — Al-Azhar University
Locations (1):
- Dental Medicine Al-Azhar University, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baccetti T, Franchi L, Cameron CG, McNamara JA Jr. Treatment timing for rapid maxillary expansion. Angle Orthod. 2001 Oct;71(5):343-50. doi: 10.1043/0003-3219(2001)0712.0.CO;2. PMID 11605867
- [Background] McNamara JA. Maxillary transverse deficiency. Am J Orthod Dentofacial Orthop. 2000 May;117(5):567-70. doi: 10.1016/s0889-5406(00)70202-2. No abstract available. PMID 10799117